CLINICAL TRIAL: NCT02854891
Title: Ambient Light Levels in the Kindergarten and Schools and the Relation to Refractive Development
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0027:16
Record Dates: First submitted 2016-03-21; First posted 2016-08-04 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-03

CONDITIONS: Myopia
Keywords: Effects; Heat; Light
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: autorefractometer, A-scan ultrasound — A measurement of refraction will be made by the Autorefractometer. A measurement of the eyes' biometer data will be made by A-scan ultrasound.

SUMMARY:
Myopia, the most common human eye disorder, is a phenomenon characterized by an unconstrained elongation of the eye globe There are number of theories concerning the environmental effect on the emmetropization process, most are related to childhood exposure to outdoor activity, near work and sleep with night light. Studies in lab animals found an association between intensity of ambient lighting and myopia development.

In this study, the investigators will examine the ambient light in kindergarten and schools and their relation to refractive error. Diurnal luminance in kindergarten and school class room will be measured and correlated to biometric measures such as refraction, axial length and keratometry.

ELIGIBILITY:
Inclusion criteria

* Every child that have been studying in the same class for the last 6-12 months (kindergarten and school respectively).

Exclusion criteria

* Noncooperative child or parents.
* Ocular surgery.
* Ocular genetic disease.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Two hundred children at ages range from kindergarten to junior year of high-school (4-17), enrolled in the formal education system in hadera and it surrounding.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-02 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
the relation between the level of myopia and light intensity | change from baseline at the start point of the study, after 6 months and after 12 months
  an analysis of the correlation between the two variables. the data will be collected as reported in the secondary outcome measures (number 2 and 5).

SECONDARY OUTCOMES:
levels of ambient light intensity | natural light- start of study and once a month until completion, average of 1 year. artificial light- once at the start point of the study
  Classes that are influenced by sunlight will be examined for light levels at a specific day of each month . For classes that are not influenced by sunlight, light source and levels will be documented. the measurement will be held until study completion.
  will be measured by luxmeter. the results will be in LUX (standardised unit of measurement of light intensity)
measurement of axial length | change from baseline at the start point of the study, after 6 months and after 12 months
  will be measured using A-scan ultrasound. the results will be in millimeters.
measurement of Visual acuity | change from baseline at the start point of the study, after 6 months and after 12 months.
  will be measured using LogMAR chart.
measurement of refraction | change from baseline at the start point of the study, after 6 months and after 12 months.
  will be measured using autorefractometer. the results will be in diopter
measurement of cornea curvature | change from baseline at the start point of the study, after 6 months and after 12 months.
  will be measured using autorefractometer. the results will be in millimeters.

IPD SHARING:
Plan to Share IPD: Yes